CLINICAL TRIAL: NCT06875713
Title: Parenting for Lifelong Health in Kuwait (DAYEM) - a Randomized Controlled Trial
Brief Title: Parenting for Lifelong Health Program in Kuwait
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Hind Almazeedi, Head of Research Unit and Prevention Programs Unit at CPO, Ministry of Health, Kuwait
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024/2735
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Child Development; Parenting Behavior; Parenting Intervention; Child Mental Health
Keywords: Parenting interventions; positive parenting; child well-being; child maltreatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): The intervention group will participate in eight in-person sessions of the PLH program, supplemented by the use of a digital parenting program (ParentApp) aimed at enhancing positive parenting behaviours.
  Interventions: Behavioral: Parenting for Lifelong Health Program (DAYEM)
- control group (Active Comparator): The control group will receive education on adult nutrition over the same period.
  Interventions: Behavioral: Adult nutrition

INTERVENTIONS:
Behavioral: Parenting for Lifelong Health Program (DAYEM) — This intervention consists of the Parenting for Lifelong Health (PLH) program, delivered through eight in-person sessions, supplemented by a digital parenting program (ParentApp). The intervention aims to enhance positive parenting behaviors and reduce child maltreatment.
  Arms: intervention group
Behavioral: Adult nutrition — The control group will receive education on adult nutrition over the same period.
  Arms: control group

SUMMARY:
Parenting interventions play a crucial role in promoting positive parent-child interactions, which are fundamental to fostering child well-being. Over the years, substantial progress has been made in understanding the importance of these interactions, particularly in the context of early childhood development. Positive parent-child interactions lay the groundwork for various aspects of child development, including socioemotional skills, academic performance, and mental health. Evidence-based parenting programs have demonstrated strong effectiveness in promoting positive parenting and preventing child maltreatment. The Parenting for Lifelong Health (PLH) program has yielded positive outcomes in many countries. This project aims to culturally adapt the PLH program and conduct a randomized controlled trial (RCT) to assess its feasibility and effectiveness in Kuwait.

ELIGIBILITY:
Inclusion Criteria:

* A primary caregiver of children aged 2-9 years
* Over the age of 18.
* Kuwaiti
* Lives in Kuwait
* Speaks Arabic

Exclusion Criteria:

* Non-Arabic speakers
* Non-Kuwaitis
* Parent whose co-parent is participating in study
* Not resident of Kuwait
* Target child has mental disability or special needs
* Facilitator, supervisor, or caregiver contributor in the DAYEM program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Parenting and Discipline Strategies | three time points: pre-intervention, post-intervention (one week after the intervention ends ), and four months post-intervention
  This section measures the frequency of various discipline strategies used by parents or caregivers in the past 30 days (9 items), including physical (e.g., spanking, using objects, grabbing, pinching) and psychological (e.g., yelling, shaming, ignoring, threatening) disciplinary practices. Responses range from 0 time to 8/8+ times, providing insight into parenting behaviors and disciplinary approaches.

SECONDARY OUTCOMES:
Demographic and Social Information | pre-intervention
  This section measures demographic and socioeconomic characteristics, including age, gender, nationality, residence, number of children, marital and co-parenting status, education level, employment status, household income, and income satisfaction (11 items).
Child Behavioral Concerns | three time points: pre-intervention, post-intervention (one week after the intervention ends ), and four months post-intervention
  This section assesses child behavioral and emotional difficulties over the past 30 days (10 items), including irritability, anger, mood swings, defiance, dishonesty, aggression, disruptive behavior, destructiveness, cruelty, and minor theft. Responses range from 0 (Not true) to 2 (Very true), providing insight into the child's behavioral tendencies and potential conduct issues.
Parenting Experience and Well-Being | three time points: pre-intervention, post-intervention (one week after the intervention ends ), and four months post-intervention
  This section measures parenting experience and well-being by assessing the frequency of positive parenting practices over the past 30 days (10 items). It includes aspects such as quality time spent with the child, encouragement of problem-solving, engagement in fun activities, use of praise and rewards, involvement in household chores, clear communication of expectations, maintaining a calm tone, and providing explanations and preparation for challenging situations. Responses range from 1 (Never) to 7 (Most of the time), reflecting caregivers' supportive and constructive parenting behaviors.
Personal Mental Well-Being | three time points: pre-intervention, post-intervention (one week after the intervention ends ), and four months post-intervention
  This section assesses personal mental well-being over the past 30 days, measuring the frequency of positive psychological states such as optimism, sense of purpose, relaxation, problem-solving ability, mental clarity, social connectedness, and decision-making confidence (7 items). Responses range from 1 (Never) to 5 (All the time), providing insight into overall emotional resilience and well-being.
Parenting Stress and Satisfaction | three time points: pre-intervention, post-intervention (one week after the intervention ends ), and four months post-intervention
  This section measures parenting stress and satisfaction by assessing caregivers' emotional experiences and attitudes toward their parenting role. It includes aspects of happiness, closeness, enjoyment, optimism, engagement with children, feelings of being overwhelmed, and potential regrets about having children (7 items). Responses range from 1 (Strongly Disagree) to 5 (Strongly Agree), providing insight into caregivers' overall parenting experience and well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Child Protection Office - Ministry of Health, Safat, Safat, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: A promotional website for the project. — https://globalparenting.org/satellite_studies/parenting-for-lifelong-health-programme-dayem-in-kuwait-a-randomised-controlled-trial/